CLINICAL TRIAL: NCT07262749
Title: Effect of Intraperitoneal Gas Drain on Postoperative Pain After Gynecologic Laparoscopy: A Randomized Controlled Trial.
Brief Title: Intraperitoneal Gas Drainage to Reduce Postoperative Shoulder Pain After Gynecologic Laparoscopy .
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Shehata Mohamed, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IPD in gynecologic laparoscopy
Record Dates: First submitted 2025-11-21; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Shoulder Pain After Gynecologic Laparoscopy
Keywords: Laparoscopy; Shoulder Pain; Postoperative Pain; Carbon Dioxide Retention; Intraperitoneal Gas Drain; Gynecologic Surgery; Visual Analog Scale (VAS)
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative; Hypercapnia

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel groups: one receiving intraperitoneal gas drainage and one receiving standard care without drainage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraperitoneal Gas Drain (Experimental): Placement of a plastic intraperitoneal drain through the umbilical port at the end of gynecologic laparoscopy. The drain is left in place for 24 hours to facilitate passive evacuation of residual CO₂ and reduce postoperative shoulder pain.
  Interventions: Other: Intraperitoneal Gas Drain
- Standard Care (No Drain) (No Intervention): Routine postoperative care following gynecologic laparoscopy without placement of an intraperitoneal drain. Standard gas evacuation is performed at the end of the procedure.

INTERVENTIONS:
Other: Intraperitoneal Gas Drain — A plastic intraperitoneal drain is placed through the umbilical port at the end of laparoscopic surgery and left in situ for 24 hours to allow passive evacuation of carbon dioxide. This aims to reduce diaphragmatic irritation and postoperative shoulder pain.
  Arms: Intraperitoneal Gas Drain

SUMMARY:
This randomized controlled trial aims to evaluate whether the use of an intraperitoneal gas drain at the end of gynecologic laparoscopic surgery can reduce postoperative shoulder pain. Residual carbon dioxide after laparoscopy is believed to irritate the diaphragm and cause referred shoulder pain, which is a common and distressing postoperative symptom. Women undergoing gynecologic laparoscopy lasting more than 20 minutes will be randomized to receive either an intraperitoneal drain for passive gas evacuation or standard care without a drain. Shoulder pain, abdominal pain, analgesic consumption, postoperative nausea and vomiting, and recovery indicators will be assessed during the first 48 hours after surgery.

DETAILED DESCRIPTION:
Post-laparoscopic shoulder pain is a frequent complaint after gynecologic laparoscopy and is mainly attributed to residual carbon dioxide retained in the peritoneal cavity, which irritates the diaphragm and stimulates the phrenic nerve. This study is designed to investigate a simple mechanical intervention-placement of an intraperitoneal gas drain-to facilitate passive evacuation of carbon dioxide and potentially reduce postoperative pain.

Women undergoing gynecologic laparoscopy lasting more than 20 minutes at the Department of Obstetrics and Gynecology, Women's Health University Hospital, Assiut University, will be recruited and randomized into two equal groups. The intervention group will receive a plastic intraperitoneal drain placed through the umbilical port and left in situ for 24 hours postoperatively. The control group will undergo standard gas evacuation without drain placement.

Pain will be assessed using a 10-cm Visual Analog Scale (VAS) at recovery, 6, 12, 24, and 48 hours postoperatively for both shoulder and abdominal pain. Secondary outcomes include total analgesic consumption within 48 hours, incidence of postoperative nausea and vomiting, time to return of intestinal sounds, and time to first mobilization. The primary outcome is the mean shoulder pain score at 24 hours.

This trial aims to provide high-quality evidence on the effectiveness of intraperitoneal gas drainage in reducing postoperative discomfort following gynecologic laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing gynecologic laparoscopy lasting more than 20 minutes.
* Able and willing to provide informed consent.

Exclusion Criteria:

* Refusal to participate.
* Patients unable to give consent or unable to participate in pain assessment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Severity of postoperative shoulder pain using the Visual Analog Scale (VAS) | At 24 hours after surgery
  Shoulder pain severity will be assessed using the Visual Analog Scale (VAS), a 10-cm scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate worse pain.

SECONDARY OUTCOMES:
Postoperative shoulder pain (VAS) at 6 hours | At 6 hours after surgery
  Pain severity will be measured using the Visual Analog Scale (VAS), a 10-cm scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate worse pain.
Postoperative shoulder pain (VAS) at 12 hours | At 12 hours after surgery
  Pain severity will be measured using the Visual Analog Scale (VAS), a 10-cm scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate worse pain.
Postoperative shoulder pain (VAS) at 24 hours | At 24 hours after surgery
  Pain severity will be measured using the Visual Analog Scale (VAS), a 10-cm scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate worse pain.
Postoperative shoulder pain (VAS) at 48 hours | At 48 hours after surgery
  Pain severity will be measured using the Visual Analog Scale (VAS), a 10-cm scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate worse pain.
Total analgesic consumption within 48 hours | Up to 48 hours after surgery
  Total amount of opioids and NSAIDs administered during the first 48 hours after surgery will be recorded.
Incidence of postoperative nausea and vomiting | Up to 48 hours after surgery
  Number of participants experiencing nausea and/or vomiting within 48 hours after surgery.
Time to return of bowel sounds | Up to 48 hours after surgery
  Time from end of surgery until the first documented return of bowel sounds.
Time to first mobilization | Up to 48 hours after surgery
  Time from end of surgery until first ambulation.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Fayek Amin Mousa, Principal Investigator — Assiut University - Faculty of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee PS, Chen CY, Wang PC, Chao KC, Hsieh CH. Shoulder pain reaches its peak at 12 hours after gynecological laparoscopic surgery and then gradually decreases. Taiwan J Obstet Gynecol. 2025;64(2):187-193. doi:10.1016/j.tjog.2025.01.010
- [Background] Olguín-Ortega A, Carrillo-Silva J, Hernández-Enríquez M, et al. Post-laparoscopic shoulder pain and strategies for prevention. Front Med. 2024;11:1347961. doi:10.3389/fmed.2024.1347961
- [Background] Abbott J, Hawe J, Srivastava P, Hunter D, Garry R. Intraperitoneal gas drain to reduce pain after laparoscopy: randomized masked trial. Obstet Gynecol. 2001 Jul;98(1):97-100. doi: 10.1016/s0029-7844(01)01383-7. PMID 11430964
- [Background] Swift G, Healey M, Varol N, Maher P, Hill D. A prospective randomised double-blind placebo controlled trial to assess whether gas drains reduce shoulder pain following gynaecological laparoscopy. Aust N Z J Obstet Gynaecol. 2002 Aug;42(3):267-70. doi: 10.1111/j.0004-8666.2002.00267.x. PMID 12230061
- [Background] Tsai HW, Chen YJ, Ho CM, Hseu SS, Chao KC, Tsai SK, Wang PH. Maneuvers to decrease laparoscopy-induced shoulder and upper abdominal pain: a randomized controlled study. Arch Surg. 2011 Dec;146(12):1360-6. doi: 10.1001/archsurg.2011.597. PMID 22184293
- [Background] Jackson SA, Laurence AS, Hill JC. Does post-laparoscopy pain relate to residual carbon dioxide? Anaesthesia. 1996 May;51(5):485-7. doi: 10.1111/j.1365-2044.1996.tb07798.x. PMID 8694166
- [Background] Alexander JI. Pain after laparoscopy. Br J Anaesth. 1997 Sep;79(3):369-78. doi: 10.1093/bja/79.3.369. No abstract available. PMID 9389858